CLINICAL TRIAL: NCT06038916
Title: Phase Ib/II Randomized, Double-blind, Placebo-controlled Evaluation of the Safety and Initial Efficacy of STSA-1002 Injection in Patients With Acute Respiratory Distress Syndrome
Brief Title: To Evaluate The Safety and Initial Efficacy of STSA-1002 Injection in Patients With Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STSA-1002-04
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-11

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo group (Placebo Comparator): Patients in this group will receive basal treatment and placebo.
  Interventions: Drug: STSA-1002 Injection Placebo
- Low dose group (Experimental): Patients in this group will receive basal treatment and placebo+ low-dose STSA-1002.
  Interventions: Drug: STSA-1002 Injection Placebo; Drug: STSA-1002 Injection
- High dose group (Experimental): Patients in this group will receive basal treatment and High-dose STSA-1002.
  Interventions: Drug: STSA-1002 Injection

INTERVENTIONS:
Drug: STSA-1002 Injection Placebo — Intravenous infusion
  Arms: Low dose group; Placebo group
Drug: STSA-1002 Injection — Intravenous infusion
  Arms: High dose group; Low dose group

SUMMARY:
To evaluate the safety and initial efficacy of STSA-1002 injection in patients with acute respiratory distress syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old≤Age≤85 years old;
2. Pathogen results indicate respiratory viral infection;
3. Acute respiratory distress syndrome (ARDS) caused by viral pneumonia;
4. In 14haode days since the onset of respiratory infective symptoms (in 12 days for non-invasive mechanical ventilation patients);
5. PaO₂/FiO₂ ≤200 mmHg based on arterial blood gas analysis prior to randomization;
6. Most recent peripheral blood lymphocyte count ≤0.8×10^9/L prior to randomization;
7. Patients (including patients' partners) has no plans for conception during the study period and within 4 months following the last dose, and agrees to use appropriate and effective contraception (e.g., birth control pills, condoms);
8. Willing to participate in the study and signs the informed consent form

Exclusion Criteria:

1. Use of ECMO before the first administration;
2. More than 48 hours of invasive mechanical ventilation prior to the first dose;
3. Based on the researchers' overall assessment, the patient's condition improved within the first 48 hours prior to the initial dosing (predictable improvement in oxygenation indicators observed within the next 48 hours);
4. Expected survival period of less than 24 hours or a history of cardiac arrest within 4 weeks prior to screening;
5. Recent history of stroke or acute coronary syndrome;
6. Diagnosed with fungal pneumonia (Aspergillus, Mucor, Cryptococcus, or Pneumocystis jirovecii pneumonia);
7. Suspected or known cytomegalovirus infection;
8. Suspected or known active tuberculosis;
9. Experienced prolonged fluid resuscitation-resistant septic shock.
10. Severe chronic respiratory failure;
11. Deemed by the investigator as difficult to wean from ventilation due to severe underlying diseases;
12. Cardiogenic pulmonary edema or congestive heart failure;
13. Liver dysfunction;
14. Severe renal impairment or long-term dialysis;
15. Immunocompromised state;
16. A Absolute neutrophil count is excessively low;
17. Severe anemia or active bleeding;
18. Poor compliance with standard treatment;
19. Pregnant or breastfeeding women;
20. Participated in a clinical trial of a new drug and received treatment within 3 months prior to screening;
21. Any condition that the investigator believes may increase the risk to the patient or interfere with the execution of the clinical trial;
22. Known allergy to any component of the investigational drug or its excipients, or a history of hypersensitivity (e.g., allergic to two or more drugs);
23. Any other disease or condition that, in the investigator's opinion, makes the patient unsuitable for participation in this study;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2023-12-09 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Clinical remission time | Baseline to Day28

SECONDARY OUTCOMES:
28-day all-cause mortality rate | Day28 after first dose
Proportion of subjects achieving clinical remission on Day 14 and Day 28 | Day14, Day28 after first dose
Changes in PaO2/FiO2 values from baseline on Day 3, 5, 7, 10, and 14 | Day3, Day5, Day7, Day10, Day14 after first dose
Change rates in PaO2/FiO2 values from baseline on Day 3, 5, 7, 10, and 14 | Day3, Day5, Day7, Day10, Day14 after first dose
Proportion of subjects with a decrease in the level of respiratory support by ≥1 grade on Day 28 | Day28 after first dose
ICU length of stay and total hospitalization time on Day 28 (V10) | Day28 after first dose
Proportion of subjects discharged from the ICU on Day 28 | Day28 after first dose
Proportion of subjects with PaO2/FiO2 > 300 mmHg on Day 28±2 (V10) | Day28 after first dose
Time without ventilator use (invasive or non-invasive) within 28 days | Day28 after first dose
Proportion of subjects alive and not receiving mechanical ventilation on Day 28 | Day28 after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, Ph.D, Principal Investigator — China-Japan Friendship Hospital
Locations (30):
- China (30):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of the Chinese People's Liberation Army Army Medical University, Chongqing, Chongqing Municipality
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Second Hospital of Hebei Medical University City:Shijiazhuang, Shijiazhuang, Hebei
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical College, Xingxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Wuhan Jinyintan Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Xiangtan Central Hospital, Xiangtan, Hunan
  - Zhongda Hospital affiliated to Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Chengdu Medical College, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No